CLINICAL TRIAL: NCT06019039
Title: The Role of Power Doppler Ultrasonography in Localization of Epidural Catheter : an Observational Prospective Study
Brief Title: Power Doppler Ultrasonography in Localization of Epidural Catheter
Status: Completed | Type: Observational
Sponsor: Yasser S Mostafa, MD (Other)
Collaborators: Fayoum University Hospital (Other)
Responsible Party: Sponsor-Investigator, Yasser S Mostafa, MD, Lecturer of anesthesia, Fayoum University Hospital
Organization: Fayoum University Hospital (Other)
Other Study IDs: m649
Record Dates: First submitted 2023-08-15; First posted 2023-08-31 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Uterine Diseases
Keywords: Power doppler ultrasonography; Epidural catheter; Hysterectomy
MeSH Terms: conditions — Uterine Diseases | interventions — Echocardiography, Doppler; Echocardiography, Doppler, Color

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epidural Ultrasound group: After placement of the epidural catheter, parasagittal and transverse views with CFD will be obtained to identify location of the catheter within the epidural space. Two levels above and below the insertion site will be used to locate the epidural catheter.
  Interventions: Drug: Normal Saline Flush; Device: Doppler

INTERVENTIONS:
Drug: Normal Saline Flush — Five milliliters of sterile saline will be administered as a flush through the needle while recording the color flow doppler images. The same procedure will be repeated with a slow injection of 5 mL of saline. The speed of injection will not be standardized.
  Other Names: 0.9% isotonic normal saline
Device: Doppler — All color flow Doppler images will be performed with a Phillips CX50 ultrasound machine using a 5.0 MHz a low frequency curvilinear US probe. A two-dimensional transverse interspinous view was used to visualize the posterior complex (ligamentum flavum, epidural space and dura). After loss of resistance to normal saline, the color flow Doppler function will be turned on to examine flow through the epidural needle tip.
  The ultrasound probe was positioned in the transverse axis slightly below the epidural needle but still in the interspinous space .
  Other Names: Color flow Doppler

SUMMARY:
Epidural anesthesia is a widely used method for pain relief which is useful in various settings. Identification of needle entry into the epidural space (EDS) is performed most using a loss of resistance (LOR) technique, which was described in 1921 by Sicard and Forestier, and has remained largely unchanged since. Hysterectomy operations anesthesia and analgesia rely heavily on proper needle placement technique. A noninvasive approach to confirm the correct position of the epidural needle prior to injection of local anesthetics into the epidural space, would thus be beneficial. Ultrasound (US) is a noninvasive approach increasingly used in anesthesia practice. The use of color flow Doppler (CFD) may further aid in defining the epidural space. The aim of current study is to detect and confirm site of epidural catheter in hysterectomy by using color flow doppler ultrasonography.

DETAILED DESCRIPTION:
This study will be performed in the Fayoum University hospital. The study design will be prospective study. A detailed informed consent will be signed by the eligible patients .

female patients who undergoing an ultrasound guided for hysterectomy will be included in this review. The ultrasound guided epidural will be used in those in which an anticipated technical difficult landmark epidural space localization will be expected. These included those patients with diagnosis of obesity, defined as Body Mass Index (BMI) ≥35 kg/m2, and lumbar scoliosis, as well as those with poorly defined surface lumbar bone anatomy.

Demographic data, intervertebral level of insertion, dermatome level, and failure rate of epidural needle placement using CFD will be noted for each patient. Operation will be obtained via spinal epidural technique.

Sterile preparation and dropping of the area will be followed by placement of a curvilinear ultrasound transducer in a sterile sheath. The ultrasound will be used to identify the interspinous space. The epidural needle will be guided with the use of ultrasound direction by the use of an out of plane technique.

A two-hand technique will be used to manipulate the needle and ultrasound probe.

A 17-G Tuohy needle (Braun Medical, Inc., Melsungen,AG, Germany) will be advanced until loss of resistance to normal saline will be attained.

Confirmation of the epidural space with the use of CFD will be then obtained after injection of up to 10 mL of normal saline through the epidural needle.

A 21-G epidural catheter (B. Braun Medical, Inc.) will be then threaded into the epidural space.

A 22G, 50mm needle (SONOTAP,Pajunk,Geisingen,Germany will be then advanced until CSF is obtained.

Use of intrathecal local anesthetic will be then used as a bolus in the spinal space.

After loss of resistance to normal saline, the CFD function will be turned on to examine flow through the epidural needle tip.

The ultrasound probe was positioned in the transverse axis slightly below the epidural needle but still in the interspinous space .

Two-dimensional (2D) ultrasound images will be initially obtained after making adjustments on the ultrasound system.

These include an appropriate scanning depth (6-12 cm), using the "penetration" or "general" frequency range and adjusting the gain or the time gate compensation to improve image resolution.

The CFD function will be then turned on and then the window will be adjusted to be centered over the area of interest. The authors will adjust color baseline to enhance the qualitative depiction of flow. The authors also increased color gain to amplify the appearance of flow changes. The color gain was adjusted to a level that provided the best image while avoiding the display of random color speckles. The orientation and tilt of the ultrasound probe will be essential for optimal visualization of the CFD pattern.

The best views were obtained while the probe was tilted upwards, parallel to the lumbar spinous process orientation, in order to avoid shadow interference cast by the spinous process bony structure. This maneuver will optimize the 2D view by minimizing the shadowing caused by bony structures.

The color scale will be adjusted to maximize color flow while avoiding excessive aliasing.

The best images will be best seen with a color scale on the range of 12-20 without needing to adjust the baseline.

Sample size was calculated using G-Power©️ software version 3.1.7 (Institute of experimental psychology, Heinrich Heine University, Dusseldorf, Germany).Minimal sample size of patients was (60) patients. Effect size 0.47 Depending on previous research results. Two tailed type I error 0.05 and power of 80%.

Statistical analysis will be performed using SPSS version 24.0 (IBM, Armonk, NY, USA). Data will be tested for normality using the Kolmogorov-Smirnov test. Continuous variables are presented as mean ± standard deviation (SD) or median (interquartile range) as appropriate and categorical variables are presented as number of patients (%). Parametric continuous variables will be analyzed by unpaired t-test and non-parametric continuous variables will be analyzed by Mann-Whitney U test. For categorical variables, the Chi-square (X2) test or Fisher's exact test will be used as appropriate. Two-tailed p values of 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women who will have hysterectomy operation under epidural analgesia
* Women with the epidural catheter still in place
* American Society of Anesthesiologists (ASA) physical status I, II
* Age range from 30 and 70 years.

Exclusion Criteria:

* Patient refusal
* History of allergy to one of the study drugs.
* Any contraindication to regional anesthesia such as local infection or bleeding disorders

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary gynecology and obstetric care clinic in Fayoum university hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Visualization of flow relative to the interspace insertion level by color flow Doppler | 1 minute after insertion of epidural catheter
  Yes or no

SECONDARY OUTCOMES:
Level of epidural catheter insertion | 1 minute after insertion of epidural catheter
  From Lumbar level 1 to 5
Verbal numerical rating scale | 8 hours postoperatively
  0-10 where 0: no pain and 10:worst pain
Duration of epidural analgesia | First 24 hours postoperatively.
  in hours
Incidence of patchy or asymmetric block | 15 minutes after insertion of epidural catheter
  Yes or no
Maximum upper sensory block to ice as charted by the nurse | 15 minutes after insertion of epidural catheter
  Dermatomal level thoracic level 10 up to umbilicus
Intervertebral level at which the epidural catheter is inserted | 1 minute after insertion of epidural catheter
  From Lumbar level 2-3 or 3-4

OTHER OUTCOMES:
Age | 1 hour preoperatively
  in years
Height | 1 hour preoperatively
  in meter
Weight | 1 hour preoperatively
  in kilogram
Body mass index | 1 hour preoperatively
  kilogram/square meter
Duration of surgery | Up to 5 hours
  in hours

CONTACTS AND LOCATIONS:
Overall Officials: Atef M Sayed, MD, Principal Investigator — Fayoum University; Abeer S Goda, MD, Study Director — Fayoum University
Locations (1):
- Fayoum University Hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Y, He S, Zhou S. Effect of general anesthesia combined with epidural anesthesia on circulation and stress response of patients undergoing hysterectomy. Am J Transl Res. 2021 May 15;13(5):5294-5300. eCollection 2021. PMID 34150121
- [Background] Elsharkawy H, Sonny A, Chin KJ. Localization of epidural space: A review of available technologies. J Anaesthesiol Clin Pharmacol. 2017 Jan-Mar;33(1):16-27. doi: 10.4103/0970-9185.202184. PMID 28413269
- [Background] Riveros-Perez E, Albo C, Jimenez E, Cheriyan T, Rocuts A. Color your epidural: color flow Doppler to confirm labor epidural needle position. Minerva Anestesiol. 2019 Apr;85(4):376-383. doi: 10.23736/S0375-9393.18.13175-0. Epub 2018 Nov 22. PMID 30482003